CLINICAL TRIAL: NCT07329816
Title: External, Multicentre Validation of a Machine-Learning Model to Predict Colonic Adenoma in Indian Adults-A Prospective, Observational, Multicentre Study
Brief Title: External, Multicentre Validation of a Machine-Learning Model to Predict Colonic Adenoma in Indian Adults
Status: Not yet recruiting | Type: Observational
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Mohan Ramchandani, Consultant Gastroenterology, Asian Institute of Gastroenterology, India
Other Study IDs: VALID-ADENOMA-IN
Record Dates: First submitted 2025-12-26; First posted 2026-01-09 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Colonoscopy
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single prospective observational cohort: Participants undergo standard-of-care colonoscopy
  No allocation into treatment or comparison arms
  Interventions: Procedure: Not Applicable / Observational study

INTERVENTIONS:
Procedure: Not Applicable / Observational study — No study-specific intervention is administered. Participants undergo standard-of-care diagnostic colonoscopy and histopathological evaluation. A locked machine-learning model is applied to routinely collected baseline clinical and demographic data for risk prediction only, without influencing clinical management.

SUMMARY:
Colorectal adenomas are precursors to colorectal cancer (CRC). Accurate pre-procedure risk stratification could optimize colonoscopy yield and resource allocation in India, where adenoma prevalence varies by age, sex, and lifestyle/metabolic factors. ML models can integrate multiple predictors to estimate individualized risk.

Existing risk scores are largely Western; performance and calibration may not be appropriate in Indian populations with different socio-demographic and metabolic profiles. External, prospective, multicentre validation is essential before clinical implementation.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years undergoing diagnostic colonoscopy.
* Adequate bowel preparation (Boston Bowel Preparation Scale total ≥6 with each segment ≥2).
* Complete examination (cecal intubation; withdrawal time ≥6 min when no therapy).
* Availability of all model predictors per CRF.

Exclusion Criteria:

* • Known CRC or polyp, prior colectomy, polyposis syndromes, known IBD, or strong hereditary CRC syndromes (e.g., Lynch) if excluded in derivation.

  * Inadequate prep, incomplete colonoscopy, obstructing lesions preventing optical diagnosis beyond obstruction.
  * Emergency colonoscopies, therapeutic-only procedures without diagnostic intent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1000
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Area Under the Receiver Operating Characteristic Curve (AUROC) of the Machine Learning Model | 1 YEAR
  Area under the receiver operating characteristic curve (AUROC) of the machine learning-based prediction model for identifying the presence of histologically proven colonic adenoma

SECONDARY OUTCOMES:
Validation Performance of the Machine Learning Prediction Model | 1 YEAR
  Validation performance of the machine learning model for predicting colonic adenoma, assessed using AUROC, calibration metrics (Brier score), and calibration plots in an independent validation cohort.

IPD SHARING:
Plan to Share IPD: No